CLINICAL TRIAL: NCT03128463
Title: Pharmacogenomic Study on Anti-VEGF Medicine in Treatment of Macular Neovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xun Xu (Other)
Collaborators: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Peking University (Other); Air Force Military Medical University, China (Other); Tianjin Medical University (Other)
Responsible Party: Sponsor-Investigator, Xun Xu, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: 2016YFC0904800
Record Dates: First submitted 2017-03-09; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Age-Related Macular Degeneration; Polypoidal Choroidal Vasculopathy; Pathological Myopia; Conbercept; Pharmacogenomic
Keywords: Age-Related Macular Degeneration; Polypoidal Choroidal Vasculopathy; Pathological Myopia; Conbercept
MeSH Terms: conditions — Macular Degeneration; Polypoidal Choroidal Vasculopathy; Myopia, Degenerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- significantly effective group: visual improvement ≥15 letters in Early Treatment Diabetic Retinopathy Study (EDTRS) table after intravitreal injection of conbercept
  Interventions: Drug: Intravitreal injection of conbercept
- effective group: visual improvement ≥5 letters and <15 letters in EDTRS table after intravitreal injection of conbercept
  Interventions: Drug: Intravitreal injection of conbercept
- invalid group: visual improvement <5 letters and visual reduction<5 letters in EDTRS table after intravitreal injection of Combercept
  Interventions: Drug: Intravitreal injection of conbercept
- deterioration group: visual reduction≥5 letters in EDTRS table after intravitreal injection of conbercept
  Interventions: Drug: Intravitreal injection of conbercept

INTERVENTIONS:
Drug: Intravitreal injection of conbercept — We observe and collect patients with macular neovascular diseases who had intravitreal injections of conbercept. We do not interfere patients' treatment plan.

SUMMARY:
Macular neovascular diseases including age-related macular degeneration (AMD), polypoidal choroidal vasculopathy (PCV), pathological myopia (PM) and etc. can cause severe vision loss. It has become the focus of World Health Organization's blindness- prevention cause. A new anti-VEGF drug conbercept has been approved and showed good efficacy and safety in clinical trials. But the exact therapeutic regimen and the efficacy in the real world still needs to be further studied, the reasons are as follows:

1. The efficacy and safety data of conbercept are collected from rigorous random controlled trials (RCT) , it can not fully reflect the clinical application of conbercept in the real world . Therefore, the knowledge of the therapeutic regimen, safety and efficacy of conbercept is still limited.
2. Conbercept has been approved for wet-AMD only, but in clinical practice, some doctors applied other "off-label use" of conbercept. These "off-label use" has become a common phenomenon all over the world for the instruction book of drugs usually lag behind scientific researches. There is no specific law or regulatory document of drug off-label use in China until now.
3. Anti-VEGF drugs are expensive and often require multiple treatments, and some patients have poor or even no response to the drugs. This resulted enormous waste of medical resources. So, how to accurately find out those patients who have good response, how to develop individualized therapeutic regimen, and the response of patients in the real world need to be urgently investigated in the aspect of pharmacogenomics, and pharmacometabolomics.

Therefore, the investigators plan to carry out real-world researches of conbercept on treating macular neovascular diseases has significance and urgency.

The investigators intended to conduct a nationwide, non-intrusive, prospective, observational, and multicenter registration study to investigate the efficacy of conbercept in the real-world. And this study will explore the pharmacogenomics and pharmacometabolomics of conbercept, relationships of phenotype and the effectiveness of the drug, optimize the therapeutic regimen, then reduce the financial burden of patients and save the limited medical resources to achieve the purpose of accurate treatment.

For three unanswered questions raised in the background, the researchers carried out the following purposes:

1. Investigate the safety and efficacy of conbercept in treating neovascular macular disease in the real world.
2. Find out whether the "off-label use" of conbercept on PCV and PM have good efficacy.
3. Explore the pharmacogenomics and pharmacometabolomics of conbercept through large-sample registration study.

DETAILED DESCRIPTION:
Research Background

Macular neovascular disease, is a group of diseases with subfoveal choroidal neovascularization, including age-related macular degeneration (AMD), polypoidal choroidal vasculopathy (PCV), pathological myopia (PM) and etc. Due to the high permeability of immature blood vessel wall, consequent bleeding, and scarring，macular neovascularization often leads to severe vision loss. It has become the focus of World Health Organization's blindness- prevention cause [1]. Currently, the vascular endothelial growth factor (VEGF) has been widely recognized as an important promoter for neovascularization. And a series of large-scale clinical studies revealed that anti- VEGF drug is the only effective way for macular neovascular disease [2], Anti-VEGF drug has been awarded as one of the top ten scientific and technological progress by Nature magazine.

Conbercept is an anti-VEGF drug developed independently by Chinese researchers in recent years, it competitively prevents the binding of VEGF to its receptor and inhibits the downstream pathway activation, and has a higher binding affinity to VEGFA than other widely used anti-VEGF drugs. Many multicenter double blind random controlled study showed that conbercept has good efficacy and safety in treating macular neovascular diseases. In 2013, conbercept has been approved by the State Food and Drug Regulatory Administration of China and now has been widely used and recognized.

Clinical trial results showed that the conbercept has good efficacy and safety in treating macular neovascular diseases [3], but the exact therapeutic regimen and the efficacy in the real world still needs to be further studied, the reasons are as follows:

1. The efficacy and safety data of conbercept are collected from rigorous random controlled trials (RCT), it cannot fully reflect the clinical application of conbercept in the real world. Therefore, the knowledge of the therapeutic regimen, safety and efficacy of conbercept is still limited.
2. Conbercept has been approved for wet-AMD only, but in clinical practice, some doctors applied other "off-label use" of conbercept. These "off-label use" has become a common phenomenon all over the world for the instruction book of drugs usually lag behind scientific researches. There is no specific law or regulatory document of drug off-label use in China until now.
3. Anti-VEGF drugs are expensive and often require multiple treatments, besides, some patients have poor or even no response to the drugs. This resulted enormous waste of medical resources. So, how to accurately find out those patients who have good response, how to develop individualized therapeutic regimen, and the response of patients in the real world need to be urgently investigated in the aspect of pharmacogenomics, and pharmacometabolomics.

Therefore, the investigators plan to carry out real-world researches of conbercept on treating macular neovascular diseases has significance and urgency.

Scientific assumptions

The investigators intended to conduct a nationwide， non-intrusive, prospective, observational, and multicenter registration study to investigate the efficacy of conbercept in the real-world. And this study will explore the pharmacogenomics and pharmacometabolomics of conbercept, relationships of phenotype and the effectiveness of the drug, optimize the therapeutic regimen, then reduce the financial burden of patients and save the limited medical resources to achieve the purpose of accurate treatment.

For three unanswered questions raised in the background, the researchers carried out the following purposes:

1. Investigate the safety and efficacy of conbercept in treating neovascular macular disease in the real world.
2. Find out whether the "off-label use" of conbercept on PCV and PM have good efficacy.
3. Explore the pharmacogenomics and pharmacometabolomics of conbercept through large-sample registration study.

Research Plan

Program schedule: Total 2 years (1 year on enrollment, 1-year on observation) Start time: February of 2017 (FPFV, First Time Patient First Visit) End time: December of 2018 (LPLV, the last time Last Patient Last Visit) Clinical study report (CSR): December of 2018; Publish: June of 2019

This is an observational study, the investigators aim to observe and collect 5000 patients from forty nationwide ophthalmic centers that receive ocular injections of conbercept to treat macular neovascular diseases during December 2016- November 2017. And the follow-up observation last for one year. The investigators do not interfere patients' treatment plan during the entire research.

Registration time:

V1: baseline (enrollment period), V2: 1month after treatment, V3: 3 months, V4: 6 months, V5: 12 months.

Data collection and transfer:

In each visit, patients' demographic information, vital sign, history of systematic diseases, concomitant medication, eye disease history, eye examinations record, safety information and blood samples are collected. Clinical data and fundus imaging data collected by forty clinical centers will be uploaded to Shanghai Jiaotong University Ophthalmic Reading Center database then be analyzed and evaluated together.

Statistics Program: Statistical general principles:

All data will undergo descriptive statistics and statistical tests，analysis will be based on baseline and follow-up data.

Sample size:

Plan to enroll 5,000 patients by 40 hospitals. The amount will depend on the registration capacity and follow-up rate.

Safety: observe the number of cases and the percentage of adverse events and severe adverse events of conbercept in real world.

Possible bias and solutions:

Patients lost to follow (such as patients from other places, can not undergo regular local follow up): Solution 1, enroll in local patients or patients who plan to have regular and long-term follow-up in our hospital; 2, Follow up and register by telephone.

Poor patient compliance: offer some compensation for patients' transport costs.

Patients who cannot afford the drugs due to economic conditions: pharmaceutical has policies on drug donation for this population.

Quality control and Management:

Object Data Management: Ensure that all enrolled patients have signed informed consent. Each visit information should be timely, accurately and completely recorded and entered into the electronic case report form (CRF). The electronic CRF should be consistent with the original medical records. All adverse events, concomitant medications should be documented, serious adverse events should be reported to the relevant authorities within 24 hours.

Follow-up management: follow-up should be conducted according to required time point and rules. Researchers should try to find out the reasons of losing visit and avoid them. If patients failed to come to clinic, then the researchers should make a phone call follow up. If patients refused to continue participating in the study for some concerns, they should be interpreted by reasonable encourages to continue cooperation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patients were diagnosed with macular neovascular disease (wet age- related macular degeneration (AMD), polypoidal choroidal vasculopathy (PCV)and choroidal neovascularization secondary to pathological myopia (PM) ), no gender requirement, age ≥ 18years
3. Patients plan to receive intravitreal injection of conbercept;
4. Patients should be resident in this region or who plans a long-term follow- up in the clinical center.

Exclusion Criteria:

1. Participate in other intervention therapy at the same time
2. Received anti- VEGF treatment (including intravitreal injection or systematic application) within three months prior to enrollment .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to observe and collect patients with macular neovascular diseases and are going to receive conbercept treatment. The investigators do not interfere patients's treatment plan.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
visual improvement after intravitreal injection of conbercept | Feb. 2017-Dec.2018
  The efficacy was graded as significantly effective (visual improvement ≥15 letters in EDTRS )，effective (visual improvement ≥5 letters and <15 letters in EDTRS），invalid（visual improvement <5 letters and visual reduction<5 letters in EDTRS， deterioration （visual reduction≥5 letters in EDTRS. The number and ratio of the above-mentioned grade are to be analyzed.

SECONDARY OUTCOMES:
The off-label use of conbercept in real world. | Feb. 2017-Dec.2018
  Calculate the number of cases and percentage of off-label use（%）in real world.
The application of off-label use on targeted diseases | Feb. 2017-Dec.2018
  Record the name of diseases when off-label use is applied.
The number and percentage（%）of each target diseases in off-label use. | Feb. 2017-Dec.2018
  Calculate the the number and percentage（%）of each target diseases in off-label use respectively.
The improvement of retinal edema after using conbercept | Feb. 2017-Dec.2018
  The improvement of retinal edema after using conbercept and compare the difference between central foveal retinal thickness (CRT in μm) and the baseline after 1 month, 3 months, 6 months, and 12 months.
The different therapeutic regimens | Feb. 2017-Dec.2018
  The different therapeutic regimens when conbercept is applied on different diseases in real world, including number of treatments, frequency of injection（times per year), interval time(months).
Dropout rate of the study. | Feb. 2017-Dec.2018
  Calculate the dropout rate（%) of each follow-up time and during the whole follow-up.
Predict patients' response to conbercept on treating macular neovascular diseases by analyzing macular leakage area | Feb. 2017-Dec.2018
  After 3 months treatment, compare the macular leakage area (mm2) to baseline in Fluorescein Fundus Angiography (FFA) on patients who response to conbercept treatment and patients with no response, to further analyze the potential relationship with the response / non-response.
Predict patients' response to conbercept on treating macular neovascular diseases by analyzing CNV area | Feb. 2017-Dec.2018
  After 3 months treatment, compare the CNV area (mm2) to baseline in FFA on patients who response to conbercept treatment and patients with no response, to further analyze the potential relationship with the response / non-response.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Shi, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong CW, Yanagi Y, Lee WK, Ogura Y, Yeo I, Wong TY, Cheung CMG. Age-related macular degeneration and polypoidal choroidal vasculopathy in Asians. Prog Retin Eye Res. 2016 Jul;53:107-139. doi: 10.1016/j.preteyeres.2016.04.002. Epub 2016 Apr 14. PMID 27094371
- [Background] CATT Research Group; Martin DF, Maguire MG, Ying GS, Grunwald JE, Fine SL, Jaffe GJ. Ranibizumab and bevacizumab for neovascular age-related macular degeneration. N Engl J Med. 2011 May 19;364(20):1897-908. doi: 10.1056/NEJMoa1102673. Epub 2011 Apr 28. PMID 21526923
- [Background] Li X, Xu G, Wang Y, Xu X, Liu X, Tang S, Zhang F, Zhang J, Tang L, Wu Q, Luo D, Ke X; AURORA Study Group. Safety and efficacy of conbercept in neovascular age-related macular degeneration: results from a 12-month randomized phase 2 study: AURORA study. Ophthalmology. 2014 Sep;121(9):1740-7. doi: 10.1016/j.ophtha.2014.03.026. Epub 2014 May 1. PMID 24793528
- [Background] Amoaku WM, Chakravarthy U, Gale R, Gavin M, Ghanchi F, Gibson J, Harding S, Johnston RL, Kelly SP, Lotery A, Mahmood S, Menon G, Sivaprasad S, Talks J, Tufail A, Yang Y. Defining response to anti-VEGF therapies in neovascular AMD. Eye (Lond). 2015 Jun;29(6):721-31. doi: 10.1038/eye.2015.48. Epub 2015 Apr 17. PMID 25882328
- [Derived] Qu Y, Liu Y, Fang J, Chen C, Cheng L, Xu X, Jin J, Chen X, Niu T, Wang H, Xing X, Shi X, Shen Y, Liu K. Dysregulated serum lipid profiles in neovascular age-related macular degeneration revealed by UPLC-MS/MS lipidomics. Lipids Health Dis. 2025 Sep 29;24(1):302. doi: 10.1186/s12944-025-02735-y. PMID 41023746
- [Derived] Jing J, Yinchen S, Xia C, Jing W, Chong C, Xun X, Hengye H, Kun L. Pharmacogenomic study on anti-VEGF medicine in treatment of macular Neovascular diseases: a study protocol for a prospective observational study. BMC Ophthalmol. 2018 Jul 24;18(1):181. doi: 10.1186/s12886-018-0812-4. PMID 30041608